CLINICAL TRIAL: NCT03084510
Title: REPRISE China: REpositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of Lotus Edge™ Valve System - Clinical Evaluation in China
Brief Title: REPRISE China - Clinical Evaluation in China
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study device was recalled.
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S6071
Record Dates: First submitted 2016-10-19; First posted 2017-03-21 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Stenoses, Aortic Valve
Keywords: High risk for surgical valve replacement; transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lotus Edge™ Valve System (Experimental): The Lotus Edge™ Valve System is intended to improve the aortic valve function for symptomatic patients with severe calcific aortic stenosis (aortic valve area [AVA] of <1.0 cm2 or index of <0.6 cm2/m2) who are at high risk for standard surgical valve replacement.
  Interventions: Device: Lotus Edge™ Valve System

INTERVENTIONS:
Device: Lotus Edge™ Valve System — • The Lotus Edge™ Valve System consisting of two main components:
  * a bioprosthetic bovine pericardial aortic valve, and
  * a delivery system Device sizes include 23 mm, 25 mm and 27 mm diameter.

SUMMARY:
To evaluate the safety and effectiveness of the Lotus Edge™ Valve System for transcatheter aortic valve replacement (TAVR) in symptomatic Chinese patients with calcific, severe native aortic stenosis who are considered at high risk for surgical valve replacement.

DETAILED DESCRIPTION:
1. A independent Clinical Events Committee (CEC) will adjudge the safety endpoint.
2. Subject has a documented aortic annulus size of ≥20 mm and ≤27 mm based on the center's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]).
3. Monitor will review the source data regularly to compare the EDC to ensure the data entry can be accuracy, completeness, or representativeness.
4. Will recruit maximum 62 subjects in maximum 6 sites
5. Boston Scientific's Standard Operating Procedures to address operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years.
* Subject has documented calcific, severe native aortic stenosis with an initial AVA of <1.0 cm2 (or AVA index of <0.6 cm2/m2), and a mean pressure gradient ≥40 mm Hg or jet velocity ≥4.0 m/s or doppler velocity index ≤0.25, as measured by echocardiography and/or invasive hemodynamics.
* Subject has a documented aortic annulus size of ≥20 mm and ≤27 mm based on the center's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]).
* Subject has symptomatic aortic valve stenosis with NYHA Functional Class ≥ II.
* There is agreement by the heart team (which must include a site investigator interventionalist and a site investigator cardiac surgeon) that subject is at high operative risk for surgical valve replacement (see note below for definition of high risk, the required level of surgical assessment, and CRC confirmation) and that TAVR is appropriate. Additionally, subject has at least one of the following.

  * Society of Thoracic Surgeons (STS) score ≥ 8% -OR-
  * If STS < 8%, subject has at least one of the following conditions:

    * Hostile chest
    * Porcelain aorta
    * Severe pulmonary hypertension (> 60 mmHg)
    * Prior chest radiation therapy
    * Coronary artery bypass graft(s) at risk with re-operation
    * Severe lung disease (need for supplemental oxygen, FEV1 < 50% of predicted, DLCO < 60%, or other evidence of severe pulmonary dysfunction)
    * Neuromuscular disease that creates risk for mechanical ventilation or rehabilitation after surgical aortic valve replacement
    * Orthopedic disease that creates risk for rehabilitation after surgical aortic valve replacement
    * Childs Class A or B liver disease (subjects with Childs Class C disease are not eligible for inclusion in this trial)
    * Frailty as indicated by at least one of the following: 5-meter walk > 6 seconds, Katz ADL score of 3/6 or less, body mass index < 21, wheelchair bound, unable to live independently
    * Age ≥ 90 years
    * Other evidence that subject is at high risk for surgical valve replacement (CRC must confirm agreement with site heart team that subject meets high risk definition)
* Heart team (which must include a cardiac interventionalist and an experienced cardiac surgeon) assessment that the subject is likely to benefit from valve replacement.
* Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent
* Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion Criteria:

* Subject has a congenital unicuspid aortic valve or Sievers Type 2 bicuspid aortic valve.
* Subject has had an acute myocardial infarction within 30 days prior to the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin elevation).
* Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months prior to study enrollment.
* Subject has end-stage renal disease or has serum creatinine > 3mg/dl or has creatinine clearance rate <45ml/min.
* Subject has a pre-existing prosthetic aortic or mitral valve.
* Subject has severe (4+) aortic, tricuspid, or mitral regurgitation.
* Subject has a need for emergency surgery for any reason.
* Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis.
* Subject has echocardiographic evidence of new intra-cardiac vegetation or intraventricular or paravalvular thrombus requiring intervention.
* Subject has platelet count < 50,000 cells/mm3 (50×109/L) or > 700,000 cells/mm3 (700×109/L), or white blood cell count < 1,000 cells/mm3 (1×109/L).
* Subject requires chronic anticoagulation therapy after the implant procedure and cannot be treated with warfarin (other anticoagulants are not permitted in the first month) for at least 1 month concomitant with either aspirin or clopidogrel.
* Subject has had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months, or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen, or will refuse transfusions
* Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all P2Y12 inhibitors, heparin, nickel, tantalum, titanium, or polyurethanes
* Subject has a life expectancy of less than 12 months due to non-cardiac, comorbid conditions based on the assessment of the investigator at the time of enrollment
* Subject has hypertrophic obstructive cardiomyopathy
* Subject has any therapeutic invasive cardiac or vascular procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty or pacemaker implantation, which is allowed)
* Subject has untreated coronary artery disease, which in the opinion of the treating physician is clinically significant and requires revascularization
* Subject has severe left ventricular dysfunction with ejection fraction < 20%
* Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices
* Subject has severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely, marked tortuosity, significant narrowing of the abdominal aorta, severe unfolding of the thoracic aorta, or symptomatic carotid or vertebral disease)
* Subject has thick (> 5 mm) protruding or ulcerated atheroma in the aortic arch
* Subject has an enlarged ascending aorta with the diameter > 50mm
* Subject has arterial access that is not acceptable for the study device delivery system as defined in the device Instructions For Use
* Subject has current problems with substance abuse (e.g., alcohol, etc.)
* Subject is participating in another investigational drug or device study that has not reached its primary endpoint
* Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation. Enrollment is permissible after permanent pacemaker implantation
* Subject has severe incapacitating dementia

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Through 30 days post index procedure
  All-cause mortality through 30 days post index procedure.
Mean aortic valve pressure gradient | At 30 days post index procedure
  Mean aortic valve pressure gradient at 30 days post index procedure.

OTHER OUTCOMES:
Safety endpoints adjudicated by an independent Clinical Events Committee (CEC) | peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 , 12, 24, 36, 48 & 60 months post index procedure
  Mortality: all-cause, cardiovascular, and non-cardiovascular Stroke: disabling and non-disabling Myocardial infarction (MI): periprocedural (≤72 hours post index procedure) and spontaneous (>72 hours post index procedure) Bleeding: life-threatening (or disabling) and major Acute kidney injury (≤7 days post index procedure): based on the AKIN System Stage 3 (including renal replacement therapy) or Stage 2 Major vascular complication Repeat procedure for valve-related dysfunction (surgical or interventional therapy) Hospitalization for valve-related symptoms or worsening congestive heart failure (NYHA class III or IV)
Device Performance | peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 , 12, 24, 36, 48 & 60 months post index procedure
  Successful vascular access, delivery and deployment of the study valve, and successful retrieval of the delivery system Successful retrieval of the study valve if retrieval is attempted Successful repositioning of the study valve if repositioning is attempted Grade of aortic valve regurgitation: paravalvular, central, and combined
Procedural success | peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 , 12, 24, 36, 48 & 60 months post index procedure
  device and/or procedure related serious adverse events (SAEs) and death, correct positioning of a single transcatheter valve into the proper anatomical location, intended performance of the study device (effective orifice area [EOA] >0.9 cm2 for BSA <1.6 m2 and EOA >1.1 cm2 for BSA ≥1.6 m2 plus either a mean aortic valve gradient <20 mm Hg or a peak velocity <3m/sec, and no moderate or severe prosthetic valve aortic regurgitation) at discharge or 7 days post-procedure (whichever comes first)
prosthetic aortic valve performance as measured by transthoracic echocardiography (TTE) | peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 , 12, 24, 36, 48 & 60 months post index procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
New York Heart Association (NYHA) | peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 , 12, 24, 36, 48 & 60 months post index procedure
  New York Heart Association (NYHA) functional classification
Paravalvular aortic regurgitation | At 30 days and 12 months
  Moderate or greater paravalvular aortic regurgitation (based on core lab assessment) at 30 days and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Runlin GAO, Doctor, Principal Investigator — Cardiovascular Institute and Fu Wai Hospital
Locations (1):
- Cardiovascular Institute and Fu Wai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vahanian A, Baumgartner H, Bax J, Butchart E, Dion R, Filippatos G, Flachskampf F, Hall R, Iung B, Kasprzak J, Nataf P, Tornos P, Torracca L, Wenink A; Task Force on the Management of Valvular Hearth Disease of the European Society of Cardiology; ESC Committee for Practice Guidelines. Guidelines on the management of valvular heart disease: The Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology. Eur Heart J. 2007 Jan;28(2):230-68. doi: 10.1093/eurheartj/ehl428. Epub 2007 Jan 26. No abstract available. PMID 17259184
- [Background] Thourani VH, Myung R, Kilgo P, Thompson K, Puskas JD, Lattouf OM, Cooper WA, Vega JD, Chen EP, Guyton RA. Long-term outcomes after isolated aortic valve replacement in octogenarians: a modern perspective. Ann Thorac Surg. 2008 Nov;86(5):1458-64; discussion 1464-5. doi: 10.1016/j.athoracsur.2008.06.036. PMID 19049731
- [Background] Barreto-Filho JA, Wang Y, Dodson JA, Desai MM, Sugeng L, Geirsson A, Krumholz HM. Trends in aortic valve replacement for elderly patients in the United States, 1999-2011. JAMA. 2013 Nov 20;310(19):2078-85. doi: 10.1001/jama.2013.282437. PMID 24240935
- [Background] Iung B, Cachier A, Baron G, Messika-Zeitoun D, Delahaye F, Tornos P, Gohlke-Barwolf C, Boersma E, Ravaud P, Vahanian A. Decision-making in elderly patients with severe aortic stenosis: why are so many denied surgery? Eur Heart J. 2005 Dec;26(24):2714-20. doi: 10.1093/eurheartj/ehi471. Epub 2005 Sep 1. PMID 16141261
- [Background] Varadarajan P, Kapoor N, Bansal RC, Pai RG. Clinical profile and natural history of 453 nonsurgically managed patients with severe aortic stenosis. Ann Thorac Surg. 2006 Dec;82(6):2111-5. doi: 10.1016/j.athoracsur.2006.07.048. PMID 17126120
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Ben-Dor I, Pichard AD, Gonzalez MA, Weissman G, Li Y, Goldstein SA, Okubagzi P, Syed AI, Maluenda G, Collins SD, Delhaye C, Wakabayashi K, Gaglia MA Jr, Torguson R, Xue Z, Satler LF, Suddath WO, Kent KM, Lindsay J, Waksman R. Correlates and causes of death in patients with severe symptomatic aortic stenosis who are not eligible to participate in a clinical trial of transcatheter aortic valve implantation. Circulation. 2010 Sep 14;122(11 Suppl):S37-42. doi: 10.1161/CIRCULATIONAHA.109.926873. PMID 20837923
- [Background] Hara H, Pedersen WR, Ladich E, Mooney M, Virmani R, Nakamura M, Feldman T, Schwartz RS. Percutaneous balloon aortic valvuloplasty revisited: time for a renaissance? Circulation. 2007 Mar 27;115(12):e334-8. doi: 10.1161/CIRCULATIONAHA.106.657098. No abstract available. PMID 17389271
- [Background] Dewey TM, Brown DL, Das TS, Ryan WH, Fowler JE, Hoffman SD, Prince SL, Herbert MA, Culica D, Mack MJ. High-risk patients referred for transcatheter aortic valve implantation: management and outcomes. Ann Thorac Surg. 2008 Nov;86(5):1450-6; discussion 1456-7. doi: 10.1016/j.athoracsur.2008.07.043. PMID 19049730
- [Background] Saia F, Marrozzini C, Dall'Ara G, Russo V, Martin-Suarez S, Savini C, Ortolani P, Palmerini T, Taglieri N, Bordoni B, Pilato E, Di Bartolomeo R, Branzi A, Marzocchi A. How many patients with severe symptomatic aortic stenosis excluded for cardiac surgery are eligible for transcatheter heart valve implantation? J Cardiovasc Med (Hagerstown). 2010 Oct;11(10):727-32. doi: 10.2459/JCM.0b013e328338940f. PMID 20414120
- [Background] Thomas M. The global experience with percutaneous aortic valve replacement. JACC Cardiovasc Interv. 2010 Nov;3(11):1103-9. doi: 10.1016/j.jcin.2010.10.001. PMID 21087744
- [Background] Bourantas CV, Farooq V, Onuma Y, Piazza N, Van Mieghem NM, Serruys PW. Transcatheter aortic valve implantation: new developments and upcoming clinical trials. EuroIntervention. 2012 Sep;8(5):617-27. doi: 10.4244/EIJV8I5A94. PMID 22995089
- [Result] Lindroos M, Kupari M, Heikkila J, Tilvis R. Prevalence of aortic valve abnormalities in the elderly: an echocardiographic study of a random population sample. J Am Coll Cardiol. 1993 Apr;21(5):1220-5. doi: 10.1016/0735-1097(93)90249-z. PMID 8459080
- [Result] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Result] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Result] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Result] Brown JM, O'Brien SM, Wu C, Sikora JA, Griffith BP, Gammie JS. Isolated aortic valve replacement in North America comprising 108,687 patients in 10 years: changes in risks, valve types, and outcomes in the Society of Thoracic Surgeons National Database. J Thorac Cardiovasc Surg. 2009 Jan;137(1):82-90. doi: 10.1016/j.jtcvs.2008.08.015. PMID 19154908
- [Result] Chiam PT, Ruiz CE. Percutaneous transcatheter aortic valve implantation: Evolution of the technology. Am Heart J. 2009 Feb;157(2):229-42. doi: 10.1016/j.ahj.2008.10.003. PMID 19185629
- [Result] American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; Bonow RO, Carabello BA, Kanu C, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Lytle BW, Nishimura R, Page RL, Riegel B. ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (writing committee to revise the 1998 Guidelines for the Management of Patients With Valvular Heart Disease): developed in collaboration with the Society of Cardiovascular Anesthesiologists: endorsed by the Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. Circulation. 2006 Aug 1;114(5):e84-231. doi: 10.1161/CIRCULATIONAHA.106.176857. No abstract available. PMID 16880336
- [Result] Holmes DR Jr, Mack MJ, Kaul S, Agnihotri A, Alexander KP, Bailey SR, Calhoon JH, Carabello BA, Desai MY, Edwards FH, Francis GS, Gardner TJ, Kappetein AP, Linderbaum JA, Mukherjee C, Mukherjee D, Otto CM, Ruiz CE, Sacco RL, Smith D, Thomas JD. 2012 ACCF/AATS/SCAI/STS expert consensus document on transcatheter aortic valve replacement. J Am Coll Cardiol. 2012 Mar 27;59(13):1200-54. doi: 10.1016/j.jacc.2012.01.001. Epub 2012 Jan 31. No abstract available. PMID 22300974